CLINICAL TRIAL: NCT04545684
Title: Effects of Mental Practice on Manual Gripping Motor Function: A Randomized Controlled Trial
Brief Title: Effects of Mental Practice on Manual Gripping Motor Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Autonoma de Madrid (Other)
Collaborators: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Roy La Touche Arbizu, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: uammadrid31
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-09

CONDITIONS: Hand Grasp
Keywords: Motor imagery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental practice (Experimental)
  Interventions: Behavioral: Motor imagery
- Placebo group (Placebo Comparator)
  Interventions: Behavioral: Placebo intervention

INTERVENTIONS:
Behavioral: Motor imagery — The person will have to imagine different scenarios of manual gripping
  Arms: Mental practice
Behavioral: Placebo intervention — The placebo group will imagine a place without the presence of humans.
  Arms: Placebo group

SUMMARY:
The main objective is to evaluate and quantify the manual gripping force caused by mental practice

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60
* Healthy and with no pain subjects

Exclusion Criteria:

* Any cognitive impairment that hindered viewing of audiovisual material.
* Difficulty understanding or communicating.
* Presence of systemic pathology, Central Nervous System or rheumatic disease.
* Inadequate understanding of the Spanish language to follow instructions for measuring and treatment.
* Collaboration of pregnant women.
* Underage subjects
* Subjects with pain at the time of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-30 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-02-26 (Estimated)

PRIMARY OUTCOMES:
Hand grip strength | Change from baseline and immediately post-intervention
  It is a variable of gripping force measured in the unit of Newtons
Pain pressure threshold | Change from baseline and immediately post-intervention
  Pressure Pain Threshold (PPT) is one of these tests and it is defined as the minimum force applied which induces pain. The measurement shall be carried out by using an algometer (pressure device that induces mechanical stimuli) is to standardize the amount of pressure applied in the neck region. The reliability of pressure pain thresholds according to raters or measurement frequencies is relatively high

SECONDARY OUTCOMES:
Visual and Kinesthetic Motor Imagery Ability | Immediately before the intervention
  Visual and Kinesthetic Motor Imagery Ability will be measured with Movement Imagery Questionnaire-Revised (MIQ-R). MIQ-R has four movements repeated in two subscales, a visual and a kinesthetic one. Additionally, a score between 1 and 7 is assigned, with 1 representing difficulty in picturing the motor image or difficulty in feeling the movement previously made, and 7 representing the maximum ease. The internal consistencies of the MIQ-R have been consistently adequate with Cronbach's α coefficients ranging above 0.84 for the total scale, 0.80 for de visual subscale and 0.84 for the kinesthetic subscale.
The degree of physical activity | Immediately before the intervention.
  The degree of physical activity was objectified through the The International Physical Activity Questionnaire (IPAQ) questionnaire, which allows the subjects to be divided into three groups according to their level of activity, which can be high, moderate, and low or inactive. The IPAQ consists of 7 questions about the frequency, duration and intensity of activity (moderate and intense) performed in the last seven days, as well as walking and sitting time on a workday. The IPAQ scoring protocol assigns the following MET values to walking, moderate, and vigorous intensity activity: 3.3 METs, 4.0 METs, and 8.0 METs, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU La Salle, Madrid, Spain